CLINICAL TRIAL: NCT06608979
Title: Trauma Screening/Referral and Interpersonal Violence Prevention for Women with Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016636
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Disorder; Opioid Use Disorder; Violence, Sexual; Violence, Gender-Based; Violence, Domestic
Keywords: prevention; peer support specialist; substance use disorders; posttraumatic stress disorder; interpersonal violence; intimate partner violence; sexual violence
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Opioid-Related Disorders; Coitus | interventions — Mass Screening; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Single arm design with baseline, posttest, and follow-up assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening/Referral and Prevention (Experimental): Participants will receive a brief PTSD screening, warm handoff to trauma-focused resources if screening positive, and two session peer support specialist-delivered educational program on interpersonal violence prevention.
  Interventions: Behavioral: Screening/Referral and Prevention

INTERVENTIONS:
Behavioral: Screening/Referral and Prevention — Session 1: One hour PTSD Screening/referral and Psychoeducation on interpersonal violence (consent, drug-and-alcohol-facilitated assault, intimate partner violence); Session 2: One hour sessions on Protective Behavioral Strategies for interpersonal violence (skills training)

SUMMARY:
The purpose of this project is to implement a pilot study to investigate the feasibility and preliminary efficacy of a peer support specialist delivered violence prevention program for women in substance use treatment. The program entails a posttraumatic stress disorder (PTSD) screening, resource referral, and two session interpersonal violence prevention protocol for 60 participants. In this single arm trial, women are recruited from three substance use treatment facilities. Participants complete baseline, post-intervention, one-month, and three-month follow-up assessments. Self-report surveys assess trauma exposure, knowledge and behaviors related to interpersonal violence, and intervention engagement.

DETAILED DESCRIPTION:
The majority of women entering substance use treatment have a trauma history, placing them at risk for revictimization and substance use relapse. The purpose of this project is to implement a pilot study to investigate the feasibility and preliminary efficacy of a peer support specialist-delivered violence prevention program for women in substance use treatment. The program entails a posttraumatic stress disorder (PTSD) screening, trauma-focused resource referral, and two session interpersonal violence prevention protocol for 60 participants. In this single arm trial, women are recruited from three substance use treatment facilities. Participants complete baseline, post-intervention, one-month, and three-month follow-up assessments. Self-report surveys assess demographics, trauma and sexual assault experiences, knowledge and attitudes towards sexual and intimate partner violence, protective behavioral strategies, and intervention satisfaction and engagement.

ELIGIBILITY:
Inclusion Criteria:

1) Age 18 or higher;2) female gender identity; 3) currently engaged in substance use treatment or care (behavioral, peer support, pharmacological, medical)

-

Exclusion Criteria:

1) Non-English-speaking; 2) acute physical and medical conditions that interfere with participation in educational sessions (e.g., active psychosis, suicidality).

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant identifies as female
Enrollment: 60 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
ARC3 Consent Scale | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale assesses knowledge and attitudes towards consent in sexual situations. This is a 7-item scale with scores ranging from 7 to 35, with higher scores indicating more accurate perceptions and greater knowledge of consent (Swartout et al, 2019)
Illinois Rape Myth Acceptance Scale-Short Form | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).f
  This self-report scale assesses agreement with rape myths. We selected 10 items from the scale, with scores ranging from 10 to 70, with higher scores indicating higher agreement with rape myths. (Payne, Lonsway, & Fitzgerald, 1999).
Attitudes Towards Dating Violence | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale consists of 3 items assessing agreement with violence-supportive attitudes in dating situations. Scores range from 3 to 15, with higher scores indicating greater agreement with violence-supportive norms. (Price et al., 1999)
Dating Behavior Survey | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale consists of 17 items that assess perceived likelihood of engaging in protective behavioral strategies while dating. Scores range from 17 to 102, with higher scores indicating greater likelihood of engaging in protective behavioral strategies. Adapted from Breitenbecher, 2008.
Coping Responses to Sexual Aggression | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale consists of 16 items assessing perceived likelihood of engaging in various coping strategies to resist sexual aggression. Scores range from 16 to 96, with higher scores indicating higher perceived likelihood of resistance. (Macy, Nurius, & Norris, 2007).
Barriers to Resistance | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale consists of 13 items assessing perceived barriers to resisting sexual aggression. Scores range from 13 to 52, with higher scores indicating higher perceived barriers to resistance (Norris, Nurius, & Dimeff, 1996).
Knowledge and Use of Resources | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report scale assesses 1) how aware participants are of various community resources and 2) whether resources have been accessed in the past month. The first 13 item awareness subscale results in total scores ranging from 13 to 65, with higher scores indicating higher levels of awareness. The second subscale results in scores ranging from 0 to 13, with higher scores indicating more resources accessed.

SECONDARY OUTCOMES:
Sexual Experiences Survey Short Form Victimization | Participants complete this measure at baseline, 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report survey consists of 30 items assessing experiences with various forms of sexual victimization over the past three months. Scores range from 0 to 30, with higher scores indicating more types of sexual victimization experiences endorsed.(Koss et al., 2007)
PC-PTSD-5 | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report survey assesses past month posttraumatic stress disorder symptoms with 5 screener items. Scores range from 0 to 5, with higher scores inidicating higher likelihood of meeting criteria for PTSD.
PHQ-2 (Depression) | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report survey consists of two depression screener items, with scores ranging from 0 to 6. Higher scores indicate higher likelihood of meeting criteria for major depressive episode over the last two weeks.
CAGE-AID (Substance Use) | Participants complete this measure at baseline, post intervention (2 weeks), 1 month follow-up (6 weeks), and 3 month follow-up (18 weeks).
  This self-report inventory assesses past three month symptoms of substance use disorders with 4 items. Scores range from 0 to 4, with higher scores indicating higher likelihood of meeting criteria for a current substance use disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Zinzow, Ph.D., Principal Investigator — Clemson University
Locations (2):
- United States (2):
  - Addiction Medicine Clinic, Prisma Health Upstate, Greenville, South Carolina
  - The Phoenix Center, Greenville, South Carolina

REFERENCES:
- [Derived] Zinzow HM, Pericot-Valverde I, Smalls L, Brancato MG, Chapman G, Smith A, Thompson A, Greco C, Shank M, Eichelberger KY, Smith K, Litwin AH. A Peer Support Specialist-Delivered Sexual and Intimate Partner Violence Prevention Program for Women in Substance Use Treatment: Protocol for a Single-Arm Trial. JMIR Res Protoc. 2025 Aug 8;14:e68673. doi: 10.2196/68673. PMID 40779309